CLINICAL TRIAL: NCT06980844
Title: Interpretation of the Role of Eosinophils in Diffuse Interstitial Pneumopathies
Acronym: INTREPID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022_0155
Record Dates: First submitted 2025-04-09; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease
Keywords: T2 response; Eosinophil; Pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Patients with diffuse interstitial lung disease with eosinophilic polymorphonuclear cell > 300/mm3 in blood (ILD-eosinophilic polymorphonuclear cell group of interest) and eosinophilic polymorphonuclear cell < 100/mm3 in blood (ILD non-eosinophilic polymorphonuclear cell control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILDs eosinophilic polymorphonuclear cell (Other): Patients with diffuse interstitial lung disease with eosinophilic polymorphonuclear cell > 300/mm3 in blood (ILDs-eosinophilic polymorphonuclear cell group of interest)
  Interventions: Other: No intervention: no treatment
- ILDs NO eosinophilic polymorphonuclear cell (Other): eosinophilic polymorphonuclear cell < 100/mm3 in blood (ILDs non-eosinophilic polymorphonuclear cell control group)
  Interventions: Other: No intervention: no treatment

INTERVENTIONS:
Other: No intervention: no treatment — translationnal study: Only blood sampling and imaging will be performed on two groups of ILD patients.
  Other Names: No intervention

SUMMARY:
Diffuse interstitial lung diseases (ILDs) represent a group of rare, heterogeneous disorders of various etiologies, all sharing a common histopathological feature: fibrotic remodeling of the pulmonary parenchyma induced by a chronic inflammatory process. Although the prevalence of ILDs in France has recently been estimated at 19.4 per 100,000 inhabitants per year, they are frequently encountered in clinical practice due to their need for specialized hospital care. ILDs are associated with significant morbidity and a poor prognosis, despite the heavy burden of current therapeutic strategies. This highlights the urgent need to identify new therapeutic targets for these diseases.

Eosinophilic polymorphonuclear cell could represent one such target. As a source of pro-fibrotic mediators such as TGF-β, they may contribute to pulmonary fibrosis from a clinical standpoint. Our hypothesis is that a component of bronchial exacerbation in ILD patients may involve a type 2 immune response through the recruitment and activation of eosinophilic polymorphonuclear cell.

Given their role in pro-fibrotic signaling, our objective is to characterize type 2 immunity parameters-focusing in particular on eosinophilic polymorphonuclear cell-using a multi-source approach in a cohort of ILD patients. If type 2 immunity is significantly present in this population (referred to as ILD-eosinophilic polymorphonuclear cell), the investigators will investigate the role of eosinophilic polymorphonuclear cell in vitro using a co-culture model involving eosinophilic polymorphonuclear cell and respiratory epithelial cells (both bronchial and alveolar). Based on the results obtained, future prospects include evaluating the effects of biotherapy within this model as a preliminary step toward a subsequent clinical study.

DETAILED DESCRIPTION:
From a pathophysiological perspective, the development of interstitial lung disease (ILD) involves progressive inflammation and fibrosis. These processes gradually remodel the structure of the pulmonary parenchyma-comprising alveoli, alveolar ducts, and bronchioles-into fibrotic tissue. The etiology of ILDs is multifactorial: they may be genetic , environmental, or idiopathic.

Fibrosis leads to clinical symptoms such as progressively worsening dyspnea, dry cough, diffuse fine crackles on auscultation, oxygen desaturation, and general deterioration of the patient's condition. Pulmonary function tests (PFTs) typically reveal a restrictive ventilatory defect combined with impaired alveolar diffusion, indicating reduced gas exchange capacity.

Radiological findings may vary and commonly include one or more of the following: ground-glass opacities, reticulations, traction bronchiectasis, honeycombing, and septal thickening. Although high-resolution chest CT is a key tool in ILD diagnosis, histopathological examination of lung biopsies remains the gold standard. The presence of inflammatory and fibrotic tissue infiltration is the hallmark diagnostic criterion. However, this approach requires bronchoscopy and is highly invasive, particularly for frail patients.

Indeed, ILD patients are susceptible to acute exacerbations, which are characterized by sudden and severe clinical deterioration in respiratory function and can be life-threatening. This phenomenon is well-documented in idiopathic pulmonary fibrosis (IPF).

Most diagnoses are established by multidisciplinary discussion (MDD), involving specialists from various fields. While MDD provides a working diagnosis, etiological classification remains suboptimal for many interstitial diseases. For instance, distinguishing between hypersensitivity pneumonitis, IPF, and ILDs associated with rheumatoid arthritis can be challenging-even with advanced imaging techniques.

This has led to more pragmatic classifications such as progressive fibrosing interstitial lung diseases (PF-ILDs), where the focus shifts from precise etiology to the presence of a treatable fibrotic phenotype responsive to antifibrotic therapies.

When an etiological diagnosis is straightforward, treatment is targeted: immunosuppressants for connective tissue disease-related ILDs, or antifibrotic agents such as pirfenidone or nintedanib for IPF or fibrosing forms of other ILDs. Unfortunately, despite these therapies, prognosis remains poor for most ILDs-largely due to the occurrence of exacerbations, which are typically managed with high-dose corticosteroids. Over time, patients may progress to chronic respiratory failure requiring long-term oxygen therapy.

This underscores the need for novel therapeutic strategies to improve both functional status and survival.

Given the fibrotic component of the inflammatory response, one avenue of investigation is to identify the biological drivers of ILD onset from a mechanistic and functional standpoint. In this context, some studies have suggested that inflammation may involve the recruitment of eosinophilic polymorphonuclear cells (E-PMNs). While the role of E-PMNs in ILD pathogenesis has been strongly hypothesized, it has yet to be definitively demonstrated.

E-PMNs are circulating granulocytes derived from the hematopoietic lineage. Produced in the bone marrow, they are recruited into tissues following activation of the type 2 (T2) immune response, orchestrated by Th2 lymphocytes and type 2 innate lymphoid cells (ILC2), primarily via the secretion of IL-5.

This T2 response is triggered by parasitic antigens, allergens, or tissue injury. Although beneficial against parasites, eosinophil recruitment and activation are central to allergic and respiratory pathophysiology and have multiple clinical consequences. E-PMNs release pro-fibrotic mediators such as TGF-β and have been implicated in conditions like chronic eosinophilic pneumonia (Carrington disease) and even endomyocardial fibrosis.

In humans, hypereosinophilia (eosinophilic polymorphonuclear cell ≥ 1500/mm³) is a known cause of pulmonary fibrosis. However, new diagnostic thresholds are being considered, as levels ≥150 cells/mm³ may already indicate pathological eosinophilia.

Our clinical observations have revealed the coexistence of ILD and bronchial disease, as well as characteristic "bronchial-type" exacerbations in ILD patients with unexpected eosinophilia. Investigators believe that both this association and its clinical relevance are currently underestimated in the management of ILD.

There is no established consensus on the management of ILD exacerbations, which often result in short- or medium-term mortality. However, recent studies suggest that high-dose corticosteroid therapy may improve outcomes, supporting our hypothesis of a T2-driven "bronchial-like" inflammatory component in some ILD patients.

Nonetheless, corticosteroids are not always effective and may lead to significant side effects, including heightened infection risk and cardiovascular complications.

In this context, E-PMNs could represent the common pathological link between ILD and bronchial inflammation and may serve as an actionable therapeutic target. This would open the door to existing biotherapies, already available in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* PID-PNE interest group (n= 30 patients): Adult subjects followed for chronic interstitial lung disease with a follow-up duration > 1 year with at least one biological sample showing a circulating PNE level > 300/mm3 during their follow-up, without any prescription of systemic corticosteroid therapy and antifibrotic agents (PIRFENIDONE and NINTENADIB) responsible for modulation of the eosinophil count.

  15 patients followed for Idiopathic Pulmonary Fibrosis (IPF) and 15 patients with another etiology of ILD will be selected.
* PNE ILD control group (n= 30 patients): Adult subjects with ILD with a PNE level < 150/mm3 during their follow-up, without any prescription of systemic corticosteroid therapy and antifibrotic agents (PIRFENIDONE and NINTENADIB). - Have signed a consent form.
* Be affiliated with a health insurance plan.

Exclusion Criteria:

* Patients under 18 years of age
* Patients over 75 years of age
* Pregnant patients
* Subjects with eosinophilic granulomatosis with polyangiitis (Churg-Strauss)
* Subjects with hypereosinophilic syndrome (NEP > 1500/mm3)
* Subjects with chronic idiopathic eosinophilic pneumonia (Carrington disease)
* Subjects with drug-induced interstitial lung disease
* Subjects with respiratory failure (acute and chronic: SaO2 > 92% throughout the procedure)
* Subjects with unstable heart disease
* Subjects with severe comorbidities
* Subjects receiving oxygen therapy
* Subjects deprived of liberty or under guardianship -Patients subject to a guardianship and judicial safeguard measure
* PID-PNE or non-PID PNE patients receiving systemic corticosteroid therapy or antifibrotic treatment (PIRFENIDONE and NINTENADIB)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients will not be included in the study
Enrollment: 60 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2028-08-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
The highlighting of significant differences in parameters related to T2 immunity (notably eosinophilic polymorphonuclear cell) in diffuse interstitial lung disease-EPN cells patients compared to no eosinophilic polymorphonuclear cell in ILDs patients. | Two years
  T2 immunity caractirization. A description of the variables will be provided, by median and interquartile for quantitative variables, taking into account the numbers in each group, and by number and percentages for qualitative variables. Differences in variables between the two groups will be tested using the Chi-square test or Fisher's exact test for qualitative variables and the Mann-Whitney test for quantitative variables.
  To address the primary objective, variables with a p-value <0.20 will be included in the multivariate model. A forward-backward multiple logistic regression will be performed to identify predictive factors for differentiation in epithelial damage and fibrotic phenomena between the two population groups.

SECONDARY OUTCOMES:
To define whether blood eosinophilia is analogous to bronchial eosinophilia in ILDs patients | Two years
  T2 immunity caractirization
To determine whether bronchial eosinophilia is a characteristic that can be targeted by anti-T2 biotherapy | two years
  T2 immunity caractirization
validate these observations from an experimental point of view on an in vitro model of healthy epithelium in coculture with PNE from the blood of PID patients presenting with eosinophilia. | two years
  T2 immunity caractirization

CONTACTS AND LOCATIONS:
Locations (1):
- Drci Foch Hospital, Suresnes, Suresnes, France